CLINICAL TRIAL: NCT03398252
Title: Targeting Stress-Induced Alcohol Relapse Risk With Doxazosin XL
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No funding
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jin Ho Yoon, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HSC-MS-17-0678
Record Dates: First submitted 2017-11-06; First posted 2018-01-12 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Doxazosin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doxazosin XL (Experimental): Participants will receive increasing doses of doxazosin XL (0, 4, and 8 mg).
  Interventions: Drug: Doxazosin XL
- Placebo (Placebo Comparator): Participants will be randomized to receive a placebo for doxazosin XL.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxazosin XL — Participants will be randomized to receive increasing doses of doxazosin XL (0, 4, and 8 mg).
  Other Names: Cardura XL; Cardura
  Arms: Doxazosin XL
Drug: Placebo — Participants will be randomized to receive a placebo for doxazosin XL.
  Arms: Placebo

SUMMARY:
Participants (N=10/group) will consist of non-treatment seeking individuals with AUD.

Following informed consent and baseline screening, participants will partake in 3 stress induction sessions to assess their stress levels and cravings for alcohol. Participants will be randomized to receive either increasing doses of doxazosin XL (0, 4, and 8 mg) or placebo in a double-blind manner.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-5 criteria for AUD;
* Report excessive alcohol use as defined by CDC guidelines in the past month (>7 drinks/week for woman, >14 drinks/week for men, >3 drinks/occasion for women>4 drinks/occasion for men)3.

Exclusion Criteria:

* Physical dependence on alcohol assessed using the SCID and Clinical Institute Withdrawal Assessment for Alcohol (CIWAA)41.
* Presenting an Alcohol Use Disorders Inventory (AUDIT) score indicative of severe alcohol dependence (≥13 for women, ≥15 for men);
* Meeting criteria for substance use disorder on drugs other than alcohol and nicotine;
* Currently taking a prescribed psychoactive medication (e.g., atomoxetine for ADHD). In addition, exclusion for those individuals taking CYP3A4 inhibitors. Most participants will not be taking any concomitant medications (including over-the-counter supplements). For those who are taking an allowed medication, the study physician will determine if the medications are CYP3A4 inhibitors.
* Medical conditions contraindicating doxazosin XL pharmacotherapy (e.g., postural hypotension);
* Taking contraindicated medications such as blood pressure medications;
* Be pregnant, nursing, or planning on becoming pregnant during the course of the study;
* Have any other illness, condition, or use of medications, which in the opinion of the PI and/or admitting physician would preclude safe and/or successful completion of the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-12 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility as study attendance | Two weeks
  Attending sessions

SECONDARY OUTCOMES:
Stress as assessed by salivary cortisol levels | baseline
  Cortisol levels will be measured using the Cortisol ELISA Kit (Enzo Life Sciences).
Stress as assessed by salivary cortisol levels | Friday of week 1
  Cortisol levels will be measured using the Cortisol ELISA Kit (Enzo Life Sciences).
Stress as assessed by salivary cortisol levels | Friday of week 2
  Cortisol levels will be measured using the Cortisol ELISA Kit (Enzo Life Sciences).
Stress as assessed by self-report | baseline
  Self-reported stress on a questionnaire
Stress as assessed by self-report | Friday of week 1
  Self-reported stress on a questionnaire
Stress as assessed by self-report | Friday of week 2
  Self-reported stress on a questionnaire
Stress as assessed by heart rate | baseline
  Self-reported stress on a questionnaire
Stress as assessed by heart rate | Friday of week 1
  Self-reported stress on a questionnaire
Stress as assessed by heart rate | Friday of week 2
  Self-reported stress on a questionnaire
stress reactivity as assessed by increased blood pressure | baseline
  Blood pressure
stress reactivity as assessed by increased blood pressure | Friday of week 1
  Blood pressure
stress reactivity as assessed by increased blood pressure | Friday of week 2
  Blood pressure
Alcohol craving as assessed by the Penn Alcohol Craving Scale (PACS) | baseline
  The Penn Alcohol Craving Scale (PACS) is a 5 question self-report measure that assesses alcohol craving in the past week. Each question ranges from 0 (no craving) to 6 (highest craving). The total score on the scale ranges from 0 to 30, and higher scores indicate greater alcohol craving.
Alcohol craving as assessed by the Penn Alcohol Craving Scale (PACS) | Friday of week 1
  The Penn Alcohol Craving Scale (PACS) is a 5 question self-report measure that assesses alcohol craving in the past week. Each question ranges from 0 (no craving) to 6 (highest craving). The total score on the scale ranges from 0 to 30, and higher scores indicate greater alcohol craving.
Alcohol craving as assessed by the Penn Alcohol Craving Scale (PACS) | Friday of week 2
  The Penn Alcohol Craving Scale (PACS) is a 5 question self-report measure that assesses alcohol craving in the past week. Each question ranges from 0 (no craving) to 6 (highest craving). The total score on the scale ranges from 0 to 30, and higher scores indicate greater alcohol craving.
Alcohol Demand as assessed by the Brief Assessment of Alcohol Demand (BAAD) questionnaire | baseline
  Alcohol demand will be assessed via the Brief Assessment of Alcohol Demand (BAAD), a 3-item questionnaire ("If drinks were free, how many would have?", "What is the maximum total amount you would spend on drinking?"; and "What is the maximum you would pay for a single drink?").
Alcohol Demand as assessed by the Brief Assessment of Alcohol Demand (BAAD) questionnaire | Friday of week 1
  Alcohol demand will be assessed via the Brief Assessment of Alcohol Demand (BAAD), a 3-item questionnaire ("If drinks were free, how many would have?", "What is the maximum total amount you would spend on drinking?"; and "What is the maximum you would pay for a single drink?").
Alcohol Demand as assessed by the Brief Assessment of Alcohol Demand (BAAD) questionnaire | Friday of week 2
  Alcohol demand will be assessed via the Brief Assessment of Alcohol Demand (BAAD), a 3-item questionnaire ("If drinks were free, how many would have?", "What is the maximum total amount you would spend on drinking?"; and "What is the maximum you would pay for a single drink?").
Delay discounting for alcohol as assessed by a computerized task | baseline
  Delay discounting will be assessed for both money and alcohol using a computerized task at weekly clinic visits. Delays will range from 1 day to 25 years, and monetary values will range from $0 to $1,000. In the case of alcohol discounting, the unit of alcohol (e.g., bottle, shot, glass, etc.) and cost of alcohol will be individually assessed in order to present choices that are monetarily equivalent to the money discounting task.
Delay discounting for alcohol as assessed by a computerized task | Friday of week 1
  Delay discounting will be assessed for both money and alcohol using a computerized task at weekly clinic visits. Delays will range from 1 day to 25 years, and monetary values will range from $0 to $1,000. In the case of alcohol discounting, the unit of alcohol (e.g., bottle, shot, glass, etc.) and cost of alcohol will be individually assessed in order to present choices that are monetarily equivalent to the money discounting task.
Delay discounting for alcohol as assessed by a computerized task | Friday of week 2
  Delay discounting will be assessed for both money and alcohol using a computerized task at weekly clinic visits. Delays will range from 1 day to 25 years, and monetary values will range from $0 to $1,000. In the case of alcohol delay discounting, the unit of alcohol (e.g., bottle, shot, glass, etc.) and cost of alcohol will be individually assessed in order to present choices that are monetarily equivalent to the money discounting task.
Delay Discounting for money as assessed by a computerized task | baseline
  Delay discounting will be assessed for both money and alcohol using a computerized task at weekly clinic visits. Delays will range from 1 day to 25 years, and monetary values will range from $0 to $1,000.
Delay Discounting for money as assessed by a computerized task | Friday of week 1
  Delay discounting will be assessed for both money and alcohol using a computerized task at weekly clinic visits. Delays will range from 1 day to 25 years, and monetary values will range from $0 to $1,000.
Delay Discounting for money as assessed by a computerized task | Friday of week 2
  Delay discounting will be assessed for both money and alcohol using a computerized task at weekly clinic visits. Delays will range from 1 day to 25 years, and monetary values will range from $0 to $1,000.
Alcohol use as assessed by self-report | baseline
  Self-reported drinks per day for the past week
Alcohol use as assessed by self-report | Friday of week 1
  Self-reported drinks per day for the past week
Alcohol use as assessed by self-report | Friday of week 2
  Self-reported drinks per day for the past week

CONTACTS AND LOCATIONS:
Overall Officials: Jin Ho Yoon, PhD, Principal Investigator — The University of Texas Health Science Center, Houston

IPD SHARING:
Plan to Share IPD: Undecided